CLINICAL TRIAL: NCT03432052
Title: Clinical and Radiological Outcomes of Centralization as a Surgical Management for Radial Club Hand
Brief Title: Clinical and Radiological Outcomes of Centralization of Radial Club Hand
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, El-Taher Alaa Eldin Ahmed Eid, principle Iinvestigator, Assiut University
Other Study IDs: radial club hand
Record Dates: First submitted 2018-02-02; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Radial Clubhand
Keywords: centralization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: centralization — Wrist centralization involves aligning the distal ulna with the middle finger metacarpal and passing a large Kirschner wire or a small Steinmann pin through the middle finger metacarpal, carpus, and ulna for temporary stability. This is followed by soft tissue balancing in order to counteract the volar and radial directed force vectors consisting of reefing the ulnocarpal wrist capsule and transferring the extensor carpi ulnaris muscle distally and flexor carpi ulnaris muscle dorsally on the wrist.

SUMMARY:
Assess the recurrence of deformity after wrist Centralization in cases of radial club hand and effect of the procedure on the ulnar lengthening , ulnar bowing , hand function and parent satisfaction.

DETAILED DESCRIPTION:
Radial club hand is a deficiency along the radial side of the extremity. Although considerable forearm and hand anomalies are the classic findings, proximal deficiencies also can occur throughout the arm and shoulder girdle. The elbow abnormalities can include deficiences of the olecranon, capitellum, coronoid fossa, and medial epicondyle.

In 1733, Petit first described radial club hand in an autopsy of a neonate with bilateral club hands and absent radii.

Initial surgical treatment of radial club hand involved an ulnar osteotomy to correct the bow, along with splitting of the distal ulna for insertion of the carpus. Reconstruction of the radius with a bone graft to support the carpus was reported in the 1920s, and non-vascularized epiphyseal transfer was reported in 1945. Results of these procedures were disappointing. They had multiple causes of failure, including disruption of the ulnar growth plate and subsequent increase in limb-length discrepancy, inadvertent ankylosis or arthrodesis of the wrist and loss of motion, and failure of the transplanted bone to grow, with eventual loss of radial support.

Centralization of the carpus on the distal ulna has emerged as the preferred surgical technique for correcting radial clubhand.in 1893, Sayre described it consisting of seating the distal ulna into a surgically created carpal notch. Pioneers in congenital hand surgery developed the basis for this procedure. Numerous modifications have been described to obtain or maintain correction of the wrist on the ulna.

Wrist centralization involves aligning the distal ulna with the middle finger metacarpal and passing a large Kirschner wire or a a small Steinmann pin through the middle finger metacarpal , carpus ,and ulna for temporary stability. This is followed by soft tissue balancing in order to counteract the volar and radial directed force vectors consisting of reefing the ulnocarpal wrist capsule and transferring the extensor carpi ulnaris muscle distally and flexor carpi ulnaris muscle dorsally on the wrist.

ELIGIBILITY:
Inclusion Criteria:

* All patients which had done centralization in our department who are available for follow up with complete records within the past 10 years.
* Cases with radial club hand Grade 3, 4 according to Bayne-Klug classification.
* Follow up duration should be at least two years.

Exclusion Criteria:

* Patients with follow up less than 2 years.
* Cases with Radial club hand Grade 1 , 2 according to Bayne-Klug classification

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients which had done centralization in our department who are available for follow up with complete records within the past 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
recurrence of wrist deformity | at least 2 years of follow up
  HFA more than 10 degrees as Vilkki HWO severity grading for radial dysplasia consider 10 degrees is the cut-off point for mild deformity.The hand-forearm-angle (HFA) is defined as the acute intersecting angle between the longitudinal axis of the third metacarpal and a line drawn perpendicular to the distal physis of the ulna

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — http://emedicine.medscape.com/article/1243998-overview